CLINICAL TRIAL: NCT06623968
Title: A 39-year Follow-up Study on the World´s First Single Dental Implants
Status: Completed | Type: Observational
Sponsor: Branemarkkliniken (Other)
Responsible Party: Sponsor
Other Study IDs: EPN 2023-00888-01
Record Dates: First submitted 2024-09-24; First posted 2024-10-02 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Edentulism
Keywords: dental implants; edentulism
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 39 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Dental implants — Long-term follow-up study on singel-tooth implants

SUMMARY:
This is a comprehensive, long-term follow-up study of single-implant treatments. At the Brånemark Clinic in Gothenburg, Sweden, during the period of 1982-1985, 16 patients received single-tooth implants. This study evaluates the survival rate of the implants after nearly four decades, focusing on the biological and technical complications.

Of the original 16 patients with a total of 23 implants, 14 patients with 19 implants were available for the follow-up and were included in the study. Clinical and radiographic examinations were performed on these patients.

ELIGIBILITY:
Inclusion Criteria:

Patient with diagnosis singel-tooth gap Patient with singel-tooth implants

Exclusion Criteria:

patient with bridge constructions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All living patient included in the original prospective study
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 1982-12-01 (Actual); Primary Completion 1985-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Biological and technical complications | From enrollment in 1982 - today
  Long-term follow-up of singel-tooth implants with regard to biological and/or technical complications
Marginal bone level | from 1982 to today
  Marginal bone level changes in mm

IPD SHARING:
Plan to Share IPD: No